CLINICAL TRIAL: NCT02449759
Title: Evaluating Acceptance and Commitment Therapy as a Low-intensity, Manual-based, Guided Self-help Intervention for Anxiety and Depression: A Pilot Study
Brief Title: An ACT Manual-based, Guided Self-help Intervention Pilot
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 166325
Record Dates: First submitted 2015-04-29; First posted 2015-05-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT Intervention Group (Experimental): This group will receive an ACT self-help manual to be completed over the course of 6 weeks. They will also receive two brief telephone calls during the reading of the manual by a member of the research team.
  Interventions: Behavioral: ACT Intervention Group
- Control Group (No Intervention): This group will receive no intervention

INTERVENTIONS:
Behavioral: ACT Intervention Group — A six chapter, 58 page self-help manual based on the principles of Acceptance and Commitment Therapy
  Arms: ACT Intervention Group

SUMMARY:
This study aims to evaluate the effectiveness of a guided self-help intervention using Acceptance and Commitment Therapy (ACT). Half of the participants will receive the self-help manual whilst on a waiting list for individual therapy, while the other half will remain on a waiting list and not receive the manual. This study is looking specifically at individuals with mild to moderate anxiety and/or depression.

DETAILED DESCRIPTION:
Many patients are offered written self-help material as a stage 1 (low intensity) intervention for anxiety and/or depression, as recommended by the United Kingdom's National Institute for Clinical Excellence's pathways framework (http://pathways.nice.org.uk/).

Acceptance and Commitment Therapy (ACT) is an emerging therapy that has been shown to help patients with mild to moderate anxiety and/or depression in therapist-led individual and group treatments. However, few studies have shown how effective ACT is in the form of a low-intensity, guided self-help intervention.

This study seeks to find out whether an ACT-based manual, sent to patients with anxiety and/or depression, increases their ability to effectively manage their difficulties and improve their quality of life. Participants on a primary care mental health waiting list will be invited to take part in this study.

Eligible participants will be randomly allocated to one of two groups: the ACT intervention or waiting list as usual. Participants receiving the ACT intervention will be posted a manual and will be asked to read a chapter each week for six weeks. A member of the research team will also phone them on two occasions to support their use of the manual, trouble shoot any difficulties and provide encouragement. All participants will be asked to complete nine, short questionnaires sent through the post prior to and after six weeks of self-help.

By comparing the results the study will demonstrate whether the ACT intervention is effective compared to wait list as usual.

ELIGIBILITY:
Inclusion Criteria:

* On the primary care waiting list for individual therapy
* Anxiety or depression/low mood assessed using the Depression, Anxiety and Stress Scales (DASS21). Those with mild to moderate (≥ 4 and ≤ 7) mixed anxiety (including panic, agoraphobia, obsessive compulsive disorder, generalised anxiety disorder and phobias) or depressive/low mood (including dysthymia; ≥ 5 and ≤ 10) will be included.
* For those participants presenting with both anxiety and depression, at least one must reach the minimum cut off score and neither should exceed the maximum cut-off score.
* Adequate English ability
* Able to give informed consent

Exclusion Criteria:

* High suicide risk (as indicated with a risk score of >0.3 on the Clinical Outcomes in Routine Evaluation questionnaire; CORE-34
* Participants that have been flagged at the referral meeting to receive specialised individual therapy (e.g. schema-focussed therapy)
* Medication change within the last three months*
* Currently receiving or received psychological help within the last 6 months using a Cognitive Behavioural Therapy or ACT modality (e.g. Beating the Blues, Anxiety Management Groups, Mindfulness, Individual therapy)
* Currently taking part in another research study
* Intellectual impairment (e.g. a learning disability)
* Referral for a primary diagnosis, other than anxiety/depression, that would significantly over arch any work focusing on anxiety/depression even if the above criteria is met for anxiety/depression (e.g. an eating disorder whereby the stated symptoms: cognitions, physical sensations, emotions and behaviours, are orientated solely around food).

  * Those individuals who have started or changed medication within the last 3 months will still be eligible to participate, but will be put on hold until this time period has elapsed. They will be informed of this and told that they may not be entered into the trial if recruitment targets are met or individual treatment becomes available (the waiting list will be reviewed at the time).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change is being assessed using the Quality of Life BREF (WHOQOLBREF; Skevington et al., 2004) questionnaire | Baseline and 6 weeks
  26-item self-report questionnaire

SECONDARY OUTCOMES:
Change is being assessed using the Acceptance and Action Questionnaire II (AAQII; Bond, Hayes & Baer et. al, 2011). | Baseline and 6 weeks
  A 7-item, unidimensional, self-report questionnaire which measures the construct of experiential avoidance/psychological inflexibility

CONTACTS AND LOCATIONS:
Overall Officials: Shane A Ford, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Adult Psychology Department, Falkirk, Stirlingshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996